CLINICAL TRIAL: NCT03465527
Title: A Phase 2 Trial of Pre-phase Treatment Before R-CHOP Chemotherapy in Elderly Patients With Newly Diagnosed DLBCL
Brief Title: Pre-phase Treatment Before R-CHOP Chemotherapy in Elderly Patients With Newly Diagnosed DLBCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kosin University Gospel Hospital (Other)
Responsible Party: Principal Investigator, Ho Sup Lee, MD, PhD. associate professor, Division of hematology-Oncology, Kosin University Gospel Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Prephase
Record Dates: First submitted 2018-01-08; First posted 2018-03-14 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prednisolone (Experimental): Prednisolone 50mg bid po or iv (equivalent dose of other steroid) for 5 days ± 2 days
  Hydration, antibiotics, allopurinol, nutritional supplements, and so on.
  Interventions: Drug: PrednisoLONE 50 MG

INTERVENTIONS:
Drug: PrednisoLONE 50 MG — Prednisolone 50mg bid po or iv (equivalent dose of other steroid) for 5 days ± 2 days

SUMMARY:
A phase 2 trial of pre-phase treatment before R-CHOP chemotherapy in elderly patients with newly diagnosed DLBCL

DETAILED DESCRIPTION:
R-CHOP Chemotherapy Cataract treatment with anterior steroids Phenotypic effects Evaluate the felony associated with the procedure for the primary purpose. This study evaluated efficacy, treatment outcome and safety for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically the first large-scaled B-cell lymphoma patient
2. Diagnosis time 65 years old or older
3. Patients planning R-CHOP chemotherapy
4. Ann Arbor stage 2 (bulky ≥ diameter of 7cm), stage 3 or stage 4
5. The International Prognostic Index (IPI) is a high intermediate or high risk
6. Patients without prior history of lymphoma
7. The decision to participate voluntarily in this study and the written consent of the patient

Exclusion Criteria:

1. Histologic subtypes other than CD20 positive broad-band macro-B cell lymphoma
2. Large B-cell lymphoma involving the central nervous system
3. Inadequate systemic disease A. Patients with clinically significant heart disease (congestive heart failure, symptomatic coronary artery disease, cardiac arrhythmia) or myocardial infarction within the past 6 months B. Serious neurological and psychiatric illness C. Serious active infection D. Other medical illnesses other than clinical trials
4. If the drug used in this study is allergic
5. If you do not agree to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
(treatment-related mortality rate; TRM) | an average of 1 year
  treatment-related mortality rate

SECONDARY OUTCOMES:
IMWG fragility score before and after pre-phase treatment | an average of 1 year
  International Myeloma Working Group,( IMWG)
TRM and RR according to IMWG fragility score | an average of 1 year
  International Myeloma Working Group,( IMWG)
response rate; RR | an average of 1 year
  response rate
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | an average of 1 year
  safety
Incidence of neutropenic fever | an average of 1 year
  Incidence of neutropenic fever

CONTACTS AND LOCATIONS:
Locations (1):
- Kosin University Gospel Hospital, Busan, Sue-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided